CLINICAL TRIAL: NCT01389167
Title: Naltrexone and Behavioral Drug and HIV Risk Reduction Counseling in Russia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: St. Petersburg State Pavlov Medical University (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Marek Cezary Chawarski, Associate Professor, Yale University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0907005456; R01DA027405 (NIH)
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Opiate Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — vivitrol; Naltrexone; Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vivitrol + BDRC (Experimental)
  Interventions: Drug: Vivitrol; Behavioral: BDRC
- Vivitrol + Medical Management (Experimental)
  Interventions: Drug: Vivitrol; Behavioral: Medical Management
- Naltrexone (oral)+BDRC (Experimental)
  Interventions: Drug: Naltrexone (oral); Behavioral: BDRC
- Naltrexone (oral) + Medical Management (Experimental)
  Interventions: Drug: Naltrexone (oral); Behavioral: Medical Management

INTERVENTIONS:
Drug: Vivitrol — An extended release naltrexone formulation for intramuscular injection
  Arms: Vivitrol + BDRC; Vivitrol + Medical Management
Drug: Naltrexone (oral) — Naltrexone 50 mg pills, daily
  Arms: Naltrexone (oral) + Medical Management; Naltrexone (oral)+BDRC
Behavioral: BDRC — Manual-guided BDRC is a highly structured, educational, prescriptive, and individualized treatment that focuses on the patient's current problem areas that are immediately related to marinating abstinence in order to achieve sustained recovery from drugs. The primary goals of BDRC include education about the disease of opiate dependence and effective treatment approaches, skills and strategies to maintain drug abstinence following detoxification, reduction/cessation of drug and sexual behaviors associated with HIV transmission, and increased engagement in non-drug-related social interactions and pleasurable activities.
  Arms: Naltrexone (oral)+BDRC; Vivitrol + BDRC
Behavioral: Medical Management — Patient assigned to MM will receive manual-guided medically oriented counseling approximating the current standard of care provided in with NTM the Russian Federation, consisting of an initial introductory session (introduction to NMT and basic education about HIV risks) and subsequent, brief (up to 20 minutes) support and advice sessions once per month.
  Arms: Naltrexone (oral) + Medical Management; Vivitrol + Medical Management

SUMMARY:
The long-term goals of this study are to foster development and dissemination of evidence-based behavioral and pharmacological treatments to reduce HIV transmission, injection drug use (IDU), and heroin use in Russia. This study will examine the effects of combining behavioral therapy with naltrexone pharmacotherapy for the treatment of opiate dependence and reduction of HIV risks in opiate dependent individuals. Specifically the study will determine whether extended-release injection naltrexone has greater efficacy and is more cost-effective than oral naltrexone maintenance, whether behavioral drug and HIV risk reduction counseling (BDRC) combined with brief, medical management (MM) has greater efficacy and is more cost-effective than MM only, and whether particular combinations of medication formulation and counseling (MM only or MM plus BDRC) have greater efficacy or are more cost-effective than other combinations.

DETAILED DESCRIPTION:
With an estimated 1.6-4 million opiate users (majority with injection drug use (IDU)) and more than 940,000 HIV infected individuals (80% linked to IDU), the Russian Federation is facing the prospect of an explosive HIV epidemic. Currently in Russia, inpatient detoxification followed by oral naltrexone maintenance (NMT) is the only pharmacologic treatment for opiate dependence. Evidence-based counseling to reduce HIV transmission and relapse following detoxification is not widely available or routinely provided. Several considerations, including data from our preliminary studies, suggest that the efficacy of NMT may be improved by using extended-release naltrexone (XR/NTX) instead of oral naltrexone (O/NTX) and by combining NMT with behavioral drug and HIV risk reduction counseling (BDRC). BDRC may also improve medication adherence and promote behavioral change leading to reduced relapse risk, IDU, and other drug- and sex-related HIV risk behaviors. However, the efficacy and cost-effectiveness for reducing drug- and sex-related HIV risk behaviors and increasing duration of opioid abstinence of the various combinations of naltrexone formulation (O/NTX vs. XR/NTX) and counseling (MM only or combined with BDRC) have not been systematically evaluated. Consequently, we are proposing a 2x2 factorial randomized clinical trial evaluating the efficacy and cost-effectiveness of two medication formulations (O/NTX and XR/NTX) and two manual-guided counseling conditions (MM only or MM+BDRC) and the potential interactions between medications and counseling conditions. Following detoxification, opiate dependent subjects (N=320) will be randomly assigned to 6 months of treatment in one of four treatment groups: O/NTX+MM, XR/NTX+MM, O/NTX+MM+BDRC, or XR/NTX+MM+BDRC. Primary outcome measures include reductions in sex- and drug-related HIV risk behaviors, reductions in illicit opiate use, and treatment retention. Other outcome measures include reductions in frequency of opiate or other drug use, health status and healthcare utilization, criminal behavior and arrests, and improvements in vocational and family functioning and quality of life. All study participants will be assessed at baseline and monthly during the 6 month treatment phase and for 6 months following the active treatment phase. Data analyses will focus on the intention-to treat sample. The study results will allow evaluation of whether XR/NTX has superior efficacy or is more cost-effective than O/NTX, whether BDRC plus MM has superior efficacy or is more cost-effective than MM only, and whether particular combinations of medications and counseling have superior efficacy or are more cost-effective than other combinations.

ELIGIBILITY:
Inclusion Criteria:

* Detoxified volunteers seeking drug rehabilitation treatment will be eligible for the study

Exclusion Criteria:

* Current suicide or homicide risk
* Current psychotic disorder or major depression
* Inability to understand the consent form or assessments
* Pregnancy
* Acute hepatitis, liver failure, or liver enzymes greater than 3 times the upper limit of normal.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-09 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
reductions in sex- and drug-related HIV risk behaviors | every month during 6 months of active study phase and during the 6 month follow-up
reductions in illicit opiate use (maximum consecutive days of abstinence following detoxification and number of days of heroin or illicit opiate use in the past 30 days) | every month during 6 months of active study phase and during the 6 month follow-up
treatment retention (time to last clinical contact during outpatient treatment phase | 6 months

SECONDARY OUTCOMES:
reductions in illicit use of other drugs | every month during 6 months of active study phase and during the 6 month follow-up
improvements in vocational, family, social functioning, and quality of life indices | every month during 6 months of active study phase and during the 6 month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Pavlov University, Saint Petersburg, Russia

REFERENCES:
- [Derived] Kornor H, Lobmaier PPK, Kunoe N. Sustained-release naltrexone for opioid dependence. Cochrane Database Syst Rev. 2025 May 9;5(5):CD006140. doi: 10.1002/14651858.CD006140.pub3. PMID 40342086